CLINICAL TRIAL: NCT07024745
Title: PrEP US NoW: PrEP Utilization Through Increasing Social Capital Among YBMSM Networks With Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J Mugavero, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300007813; R34MH128072 (NIH)
Record Dates: First submitted 2025-05-22; First posted 2025-06-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: PrEP Uptake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Female Facilitator (Other)
  Interventions: Behavioral: Intervention Group
- Control Participants (Other)
  Interventions: Behavioral: Control (Standard treatment)
- Intervention Participants (Other)
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — The Intervention is 1) interact with the Us*Now mHealth app for 1 month; 2) participate in 4 weekly sessions with other group members and led by a Female Facilitator. Each week will cover a different topic - Week 1: Intersectional Stigma, Week 2: Sexual Health, Week 3: HIV Prevention, Week 4: Engagement in PrEP Care.
  Arms: Female Facilitator; Intervention Participants
Behavioral: Control (Standard treatment) — The Control group will be asked to interact with the Us*Now mHealth app for 1 month.
  Arms: Control Participants

SUMMARY:
This project is a randomized intervention looking at PrEP uptake among young, black men who identify as gay, bisexual, or same gender loving, utilizing black females within the community to help deliver study related topics. All participants will download the Us*Now mHealth app that was created specifically for this project. Participants randomized to the Intervention arm will interact with the Us*Now mHealth app and will be invited to attend 4 weekly sessions led by a black female facilitator where the topic are pre-selected by the study team. Participants randomized to the Control arm will interact with the Us*Now mHealth app only.

ELIGIBILITY:
Inclusion Criteria:

* Female Facilitators: 1) Black/African American; 2) age 18-80 years old; 3) Female; 4) able to lead weekly sessions with participants; 5) able to download the Us*Now mHealth app
* Participants: 1) Black/African American; 2) age 18-29 years old; 3) Male; 4) Identifies as gay, bisexual, or same gender loving; 5) able to download the Us*Now mHealth app

Exclusion Criteria:

* Female Facilitators: 1) does not identify as Black/African American; 2) not Female; 3) not able to lead the weekly sessions or attend the study training
* Participants: 1) does not identify as Black/African American; 2) age 30 years or older; 3) Identifies as Straight or Heterosexual; 4) not able to download the Us*Now mHealth app

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility and Acceptability | 6 months
  Participants will complete the Feasibility of Intervention Measure (FIM), Acceptability of Intervention Measure (AIM), and Intervention Appropriateness Measure (IAM) at T1 (1 month post Intervention) and T3 (3 month after T1) surveys. All measures are 4 questions, scaled responses from Completely Disagree to Completely Agree
Change in Social Capital and Internalized Homonegativity | 6 months
  Participants will complete the Personal Social Capital Scale and Internalized Homophobia Scale at T0 (baseline), T1 (1 month after Intervention), and T3 (3 months after T1) surveys. The Personal Social Capital Scale a 10 question measure, responses range from 1 (all/Alot) to 5 (None). The Internalized Homophobia Scale is a 12 question measure with True, False, and Don't Know responses.

SECONDARY OUTCOMES:
PrEP uptake | 6 months
  Participants will be asked if they are on PrEP at T0 (baseline), T1 (1 month after Intervention), and T3 (3 months after T1) surveys.
Change in sexual practices | 6 months
  Participants will be asked a Sexual Behavior Assessment at T0 (baseline), T1 (1 month after Intervention), and T3 (3 months after T1) surveys. This is a 4 question measure asking if they have had sex in past 3 months, and if it was condomless sex

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Sohail M, Hussen SA, Dougherty Sheff S, Mugavero M, Schneider J, Hightow-Weidman L, Turan JM, Lynam M, Elopre L. An mHealth App-Based Social Capital Intervention (PrEP US NoW) to Improve Sexual Health and Uptake of Pre-Exposure Prophylaxis Among Young, Black, Sexual Minority Men: Protocol for Intervention Development and a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 18;14:e66326. doi: 10.2196/66326. PMID 40966683